CLINICAL TRIAL: NCT01340885
Title: Cognitive Dysfunction in PD: Pathophysiology and Potential Treatments, a Pilot Study
Brief Title: Cognitive Decline in Non-demented PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jau-Shin Lou, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PANUC - Lou; 5P50NS062684-02 (NIH)
Record Dates: First submitted 2011-04-19; First posted 2011-04-25 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Parkinson's Disease
Keywords: attention; mild cognitive impairment; dementia
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Dementia | interventions — Atomoxetine Hydrochloride; Rivastigmine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- atomoxetine (Active Comparator): Strattera 10-30 mg b.i.d.
  Interventions: Drug: Strattera
- rivastigimine (Active Comparator): Exelon 1.5-4.5 mg b.i.d.
  Interventions: Drug: Exelon
- Placebo (Placebo Comparator): sugar pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Strattera — 10-30 mg b.i.d. for 6 weeks
  Other Names: atomoxetine
  Arms: atomoxetine
Drug: Exelon — 1.5-4.5 mg b.i.d. for 6 weeks
  Other Names: rivastigmine
  Arms: rivastigimine
Other: Placebo — 2-6 pills for 6 weeks
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the relationship between attention and quality of life and how rivastigmine and atomoxetine alter attention in non-demented persons with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Cognitive dysfunction can occur in early stage of Parkinson's disease (PD) and increases as PD progresses. Attention deficits in PD patients with dementia strongly predict the impairment of their daily living activities.

Previous studies have shown that atomoxetine improves PD executive dysfunction and rivastigmine improves attention deficits in PD patients with dementia without worsening the motor symptoms.

The aim of this study is to examine the effect of atomoxetine and rivastigmine on attention and quality of life in PD patients without disabling cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Respond to levodopa therapy

Exclusion Criteria:

* Dementia
* Psychiatric disorders including anxiety disorders, dissociative disorders, mood disorders, schizophrenia and related disorders, or ADD/ADHD
* Any clinically unstable disease such as cancer, HIV/AIDS, heart condition, liver disease, kidney or renal failure or others that might require hospitalization
* Evidence for another neurological disease (history of seizures, Alzheimer disease, multiple sclerosis or other movement disorders);
* Currently using any of the study drugs;
* Colorblindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Shin Lou, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study did not enroll enough subjects to reach meaningful results at the time of original conduct. While study data are/were retained per investigator responsibility, sincere attempts to access these data for retrospective analysis were unsuccessful.
Period: Overall Study
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study did not enroll enough subjects to reach meaningful results at the time of original conduct. While study data are/were retained per investigator responsibility, sincere attempts to access these data for retrospective analysis were unsuccessful.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Rivastigimine | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Attention Network Effects
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Quality of Life
Description: PDQ-39
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Stroop Color Word Test
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Fatigue
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Depression
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Daytime Sleepiness
Time Frame: 6 weeks
Population: as for baseline characteristics
Arm/Group | Atomoxetine | Rivastigimine | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Study did not enroll enough subjects to reach meaningful results at the time of original conduct. While study data are/were retained per investigator responsibility, sincere attempts to access these data for retrospective analysis were unsuccessful.
Arm/Group | Atomoxetine | Rivastigimine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study did not enroll enough subjects to reach meaningful results at the time of original conduct. While study data are/were retained per investigator responsibility, sincere attempts to access these data for retrospective analysis were unsuccessful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes